CLINICAL TRIAL: NCT04332237
Title: The Impact of Accidental Hypothermia on Mortality in Trauma Patients Overall and Patients With Traumatic Brain Injury Specifically: A Systematic Review and Meta-Analysis
Brief Title: Meta-Analysis Accidental Hypothermia in Trauma
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: SRMA hypothermia trauma
Record Dates: First submitted 2020-03-25; First posted 2020-04-02 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Hypothermia; Trauma; Brain Injuries, Traumatic; Morality
MeSH Terms: conditions — Hypothermia; Wounds and Injuries; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hypothermia group: Hypothermic trauma patients or hypothermic patients with traumatic brain injury specifically.
- Normothermia group: Normothermic trauma patients or normothermic patients with traumatic brain injury specifically.

SUMMARY:
This is a systematic literature review and meta-analysis investigating the effect of accidental hypothermia on mortality in trauma patients overall and patients with TBI specifically.

Literature search will be performed using the Ovid Medline/PubMed database. Studies comparing the effect of hypothermia vs. normothermia at hospital admission on in-hospital mortality will be included in meta-analysis.

DETAILED DESCRIPTION:
Accidental hypothermia is a known predictor for worse outcomes in trauma patients, but has not been comprehensively assessed in meta-analysis so far. The aim of this systematic review and meta-analysis is to investigate the impact of accidental hypothermia on mortality in trauma patients overall and patients with traumatic brain injury (TBI) specifically.

Literature search will be conducted using the Ovid Medline/PubMed database. The search strategy will be based on the PICOS strategy.

Scientific articles reporting (1) accidental hypothermia in trauma patients overall or patients with TBI specifically, (2) body temperature and time of measurement, and (3) the impact of accidental hypothermia on outcomes will be included in the qualitative review.

Two meta-analyses will be performed including (1) trauma patients overall and (2) patients with TBI specifically. Studies reporting in-hospital mortality of hypothermic and normothermic trauma patients overall or patients with TBI specifically, based on the temperature measured at Emergency Department admission, will be included in meta-analysis. Meta-analysis will be performed using a Mantel-Haenszel random-effects model. The estimated effect size for mortality will be reported as odds ratio (OR) and 95% confidence interval (CI) for each study as well as for the overall cohort.

ELIGIBILITY:
Inclusion criteria:

* Original scientific articles
* English language
* Study in trauma patients
* Reported body temperature and time of temperature measurement
* Reported impact of accidental hypothermia on outcomes

Exclusion criteria:

* Case reports
* Systematic reviews
* Articles on therapeutic hypothermia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Trauma patiens overall and patiens with traumatic brain injury specifically
Sampling Method: Non-Probability Sample
Enrollment: 776684 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2020-01-21 (Actual); Study Completion 2020-01-21 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality | From hospital admission to discharge, expected to be up to 4 weeks
  Death occurring during the hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Haltmeier, MD, Principal Investigator — Inselspital, Bern University Hospital
Locations (1):
- Inselspital, Bern University Hospial, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No